CLINICAL TRIAL: NCT01335386
Title: Efficacy and Safety of KLYX Versus Glycerine Enema in Chinese Patients With Constipation - a Randomised, Assessor-blind Pilot Study
Brief Title: Investigation of KLYX in Patients With Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FECN2006KLY-01
Record Dates: First submitted 2011-04-13; First posted 2011-04-14 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Glycerol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- KLYX (Experimental)
  Interventions: Drug: KLYX
- Glycerine (Active Comparator)
  Interventions: Drug: Glycerine

INTERVENTIONS:
Drug: KLYX
  Arms: KLYX
Drug: Glycerine
  Arms: Glycerine

SUMMARY:
This is a randomised, assessor-blind, multi-centre pilot study to investigate the comparative safety and efficacy of KLYX and glycerine enema in the symptomatic treatment of constipation in Chinese patients.

ELIGIBILITY:
Inclusion Criteria:

* Have signed the informed consent form and have been verbally explained the details of the trial and treatment procedures
* Ethnically Chinese
* Males or females aged between 18 and 65 years inclusive
* A history of constipation symptoms for at least 6 months fulfilling, with occurrence of two or more of the following symptoms during the 3 months before screening (the 3 months need not be consecutive):

  i. Very hard (pellet-like) and/or hard stools (Type 1 or 2 of the Bristol Stool Scale) for at least 25% of the time; or ii. Sensation of incomplete evacuation at least 25% of the time; or iii. Straining during defecation at least 25% of the time; or iv. Sensation of anorectal obstruction or blockage often during defecation at least 25% of the time; or v. Manual manoeuvres needed often to facilitate defecations (e.g. digital evacuation, support of the pelvic floor) at least 25% of the time; or vi. Fewer than 3 defecations per week.
* Patient has had no bowel movement (i.e. still constipated) two days prior randomisation.

Exclusion Criteria:

* Any disorder or laboratory result at Screening that in the judgement of the investigator that will place the subject at excessive risk if participating in a controlled study
* Clinically suspected to have colorectal cancer
* Significant gastroparesis or gastric outlet obstruction
* Hypersensitivity to sodium docusate and/or sorbitol
* Hypersensitivity to glycerine
* Pregnant or lactating women, women who intend to conceive, or women who are sexually active and capable of pregnancy who are not using a method of birth control (e.g. prescription hormonal contraceptives, intrauterine device, double-barrier method, male partner sterilization)
* Diabetic patients currently on insulin therapy
* Having participated in other clinical trial(s) within the 3 (three) months prior screening
* Unable to withdraw medications that may affect gastrointestinal motility such as prokinetics, erythromycin analogues, laxatives, etc.
* Unable to meet or perform study requirements: known or suspected inability to comply with the study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Overall efficacy of enema | immediately following enema administration

SECONDARY OUTCOMES:
Time to first bowel movement | Immediately following enema administration
Patient's overall satisfaction with enema treatment | Immediately following enema administration
Stool form after enema treatment | Immediately following enema administration

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (3):
- China (3):
  - Changhai Hospital, The Second Military Medical University, Shanghai
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai